CLINICAL TRIAL: NCT04967846
Title: How Do We Resolve the Social Dilemma? Facebook Features Use as a Moderator of Mental Health.
Brief Title: Social Media Effects on Mental Health
Status: Completed | Type: Observational
Sponsor: Yale-NUS College (Other)
Responsible Party: Sponsor
Other Study IDs: SM245864
Record Dates: First submitted 2021-06-16; First posted 2021-07-20 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Mental Health Issue; Mental Health Wellness 1; Mental Health Wellness 2; Social Media Addiction; Internet Addiction
Keywords: Social Media; Facebook; Mental Health; Wellbeing
MeSH Terms: conditions — Internet Addiction Disorder; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the last decade, research on social media and mental health has produced mixed results. Overall, the current findings suggest that the negative effects on mental health are exacerbated by longer and more frequent social media usage, whereas the positive effects are bolstered when social media is used to connect with other people.

With the largest number of global users, Facebook is the most frequently studied social media network. Over the past few years, the increasing concerns about the risks associated with Facebook have even translated to wider pop culture conversations, as exemplified by the 2020 documentary The Social Dilemma. In response, Facebook has rolled out a series of features supposed to mitigate these risks and encourage responsible social media usage. These features include activity trackers and reminders, unfollow and snooze buttons, and data sharing regulators. Currently, there is no research done to address whether (1) these features are used at all, and (2) whether they are successful in moderating the negative mental health consequences of Facebook usage.

This study seeks to address the gap in literature through a survey done on the crowdsourcing platform Amazon Mechanical Turk (MTurk).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers, aged 21 and above
* English proficiency
* Facebook users

Exclusion Criteria

* Participants below 21 years old
* Non-Facebook users

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruiting a representative sample of 740 people on the crowdsourcing platform Amazon Mechanical Turk (MTurk).
Sampling Method: Non-Probability Sample
Enrollment: 608 (Actual)
Dates: Start 2021-06-13 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-09-19 (Actual)

PRIMARY OUTCOMES:
Mental Health Scores | Once during the survey.
  Depression, Anxiety, and Stress Scale (DASS-21), (measured on a 4 point scale: min = 0, max = 3; higher scores indicating higher depression, anxiety and/or stress).

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Barsova, Principal Investigator — Yale-NUS College
Locations (1):
- Yale NUS, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Yale-NUS College regulations do not allow the sharing of private participant information.

REFERENCES:
- [Derived] Barsova T, Cheong ZG, Mak AR, Liu JC. Predicting Psychological Symptoms When Facebook's Digital Well-being Features Are Used: Cross-sectional Survey Study. JMIR Form Res. 2022 Aug 29;6(8):e39387. doi: 10.2196/39387. PMID 36036971